CLINICAL TRIAL: NCT03557255
Title: The Role of Preoperative Use of Levosimendan in Ischemic Cardiac Patients Undergoing Major Abdominal Cancer Surgeries: A Prospective Randomized Study
Brief Title: Levosimendan for Cardiac Patients Undergoing Major Abdominal Cancer Surgeries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ehab-Raafat.Levo
Record Dates: First submitted 2018-05-10; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan; Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- levosimendan (Active Comparator): Levosimendan was prepared in a concentration of 25 µg/ml and infusion was commenced at a rate of 0.1 µg/kg/minute without loading and continued for 24 hours before surgery.The dose was doubled if an increase of > 20 mmHg in systolic blood pressure (SBP) could not be obtained within 2 hours after starting the infusion. Indications for dose reduction were the development of hypotension (SBP < 80 mmHg) or tachycardia (heart rate > 120 beats/min) persisting for more than 10 minute or (premature beats in a frequency exceeding 6/min or occurrence of a significant arrhythmia occurring in runs). The infusion medication would be discontinued should such occurrences persist despite dose reduction.
  Interventions: Drug: Levosimendan
- control (Active Comparator): In the control group ,an identical saline infusion regimen was employed instead of levosimendan . Both patient and care giver were blinded for the study.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levosimendan — Preoperative 24 hours infusion of levosimendan for chronic heart failure patients prior to major abdominal cancer surgeries.
  Other Names: drug group
  Arms: levosimendan
Drug: Saline — Preoperative 24 hours infusion of normal saline for chronic heart failure patients prior to major abdominal cancer surgeries.
  Other Names: control group
  Arms: control

SUMMARY:
The objective of this pilot study is to evaluate the efficacy and safety of preoperative administration of levosimendan in patients with chronic heart failure scheduled for major abdominal cancer surgery assuming the reduction of both perioperative morbidity and mortality.

DETAILED DESCRIPTION:
Cardiac complications are one of the most common causes of perioperative morbidity and mortality in patients undergoing non-cardiac surgery. Heart failure (HF) is an established risk factor for postoperative cardiac complications and mortality. The risk for postoperative mortality following major non-cardiac surgery is twice as that of patients with coronary artery disease (CAD) without HF. HF occurs in 1% to 6% of patients after major surgery, the risk being higher, between 6% and 25%, in patients with pre-existing cardiac conditions such as CAD, prior HF or valvular heart disease.

Cardiovascular disease and cancer are among the leading causes of mortality worldwide. The number of patients presenting with both diseases concomitantly is likely to increase. Cardiac patients undergoing major abdominal cancer surgeries with substantial fluid shift, blood loss and severe hemodynamic instability are at higher risk for perioperative HF.Therefore, preoperative optimization of such patients is of paramount importance. Unfortunately, guidelines for the perioperative management and preparation of such patients have not been proposed. Besides, the prophylactic use of inotropic agents for preoperative optimization of patients at high risk for HF remains controversial owing to their potential to jeopardize the myocardial oxygen supply-demand balance or to induce dysrhythmias with an assumed higher mortality.

Levosimendan is a calcium sensitizer with a positive inotropic action that has been shown to safely improve cardiac performance and hemodynamics in HF patients without increasing the myocardial oxygen demand or causing dysrrhythmias. The perioperative use of levosimendan for optimization of patients with HF has been reported in few studies with promising results, mainly for cardiac patients undergoing cardiac surgeries. However, the role of levosimendan has not been thoroughly evaluated in patients with chronic heart failure (CHF) undergoing major cancer surgery.

The purpose of this prospective study is to evaluate the safety and efficacy of preoperative administration of levosimendan in patients with CHF scheduled for major abdominal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CHF with left ventricular ejection fraction < 35%, scheduled for major abdominal cancer surgery were eligible.
* Aged 18 to 75 years.

Exclusion criteria were :

* restrictive or obstructive cardiomyopathy.
* severe cardiac valvular disease.
* history of atrial fibrillation, ventricular tachycardia or fibrillation.
* resting systolic arterial pressure <80 mmHg.
* second or third degree atrioventricular block.
* Child-Pugh class C liver cirrhosis.
* severe renal failure (defined as creatinine clearance < 30 ml/min).
* Immediate postoperative complications such as surgical re-exploration for bleeding or suspected leak.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Changes in mechanical ventilation | Baseline and after two weeks
  The total duration of postoperative ventilation in days

SECONDARY OUTCOMES:
Changes in Ejection fraction | Baseline and after one week postoperative
  The improvement in the ejection fraction in percentage.
Changes in cardiac index | Baseline and after one week postoperative
  The improvement in Cardiac index (Liters/minute/square meter)
Changes in Stroke volume index | Baseline and after one week postoperative
  The improvement in stroke volume index(milliliters/square meter)
Patient total hospital length of stay | Baseline and after two weeks postoperative
  Total hospital length of stay in days.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the results ,conclusion and final recommendation can be shared with other researchers.